CLINICAL TRIAL: NCT06183177
Title: Improving Pain, Function and Quality of Life in End-Stage Knee Osteoarthritis: A Prospective Cohort Study of Whole-Body Vibration and Exercise as Bridging Therapies for Total Knee Replacement
Brief Title: Pain Function and QOL Undergoing Whole-Body Vibration and Exercise in End-Stage Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020.401
Record Dates: First submitted 2023-12-05; First posted 2023-12-27 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Knee Osteoarthritis; Pain, Joint
MeSH Terms: conditions — Osteoarthritis, Knee; Arthralgia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise + WBV Group (Experimental)
  Interventions: Other: Whole-Body Vibration; Other: Exercise
- Exercise Group (Active Comparator)
  Interventions: Other: Exercise
- Control Group (No Intervention)

INTERVENTIONS:
Other: Whole-Body Vibration — 10 minutes of whole-body vibration when performing semi-squatting or forward lunges (12-16 Hz, varying intensity from low to high depending on patients' tolerance
  Arms: Exercise + WBV Group
Other: Exercise — Four to five sessions of a physiotherapist-led exercise program with education talk (20 minutes), group exercises (30 minutes) and individual exercises (30 minutes) per week supplemented with home exercises
  Arms: Exercise + WBV Group; Exercise Group

SUMMARY:
Knee osteoarthritis (KOA) is a chronic progressive disease that imparts substantial socioeconomic burden to society and healthcare systems. The prevalence of KOA has dramatically risen in recent decades due to consistent increases in life expectancy, and demand for joint replacement continues to rise. Total knee replacement is indicated for end-stage KOA, as it is very effective in terms of pain relief, improvement of function, and quality of life. However, the investigators will be facing an unsustainable joint replacement burden, with significant healthcare budget and health workforce implications. To alleviate this problem, different strategies including reinforce the importance of education and exercise are included; as previous studies showed that less than 40% of patients with KOA received non-pharmacological treatment, indicating that the uptake of evidence-based guidelines in clinical practice and rehabilitation is still suboptimal. Several literatures revealed that quadriceps and hamstrings strength exercise could effectively reduce pain. It has widely accepted that patients with end stage KOA will eventually pursue total knee replacement as the only viable option, and exercise has low efficacy in reduction of pain and disability in this group of patients. So, the investigators would like to know whether exercise therapy can help severe KOA patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage knee osteoarthritis on queue for scheduling primary total knee replacement
* Completed 8-week course of physiotherapy program

Exclusion Criteria:

* TKR during the last 12 months
* Severe heart failure or neurological diseases affecting physical functions

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Numerical pain rating scale | Baseline, 8 weeks
  Pain assessment. Minimum value = 0, Maximum value = 10; the higher the score the worse the pain level
Range of motion (ROM) of the diseased knee | Baseline, 8 weeks
  Measure the angle of knee bending from straight (0 degree) to fully bended (180 degrees)
Gait analysis | Baseline, 8 weeks
  Measure the movement of legs from point A to B, measure the distance in cm between steps walking on a flat surface
Knee Society Score | Baseline, 8 weeks
  Score from 0 to 100. Lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.
Knee Society Functional Assessment | Baseline, 8 weeks
  Score from 0 to 100. Lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS)-Knee pain (KP) | Baseline, 8 weeks
  Score from 0 to 100. 0 representing extreme knee problems and 100 representing no knee problems.
Knee injury and Osteoarthritis Outcome Score (KOOS)-Other Symptoms (S) | Baseline, 8 weeks
  Score from 0 to 100. 0 representing extreme knee problems and 100 representing no knee problems.
Knee injury and Osteoarthritis Outcome Score (KOOS)- Activities of Daily Living (ADL) | Baseline, 8 weeks
  Score from 0 to 100. 0 representing extreme knee problems and 100 representing no knee problems.
Knee injury and Osteoarthritis Outcome Score (KOOS)-Sport and Recreation function | Baseline, 8 weeks
  Score from 0 to 100. 0 representing extreme knee problems and 100 representing no knee problems.
Knee injury and Osteoarthritis Outcome Score (KOOS)-knee-related Quality of Life (QOL) | Baseline, 8 weeks
  Score from 0 to 100. 0 representing extreme knee problems and 100 representing no knee problems.
Timed Up and Go test | Baseline, 8 weeks
  Score from 1 to 5. 1 indicates "normal function" and 5 indicates "severely abnormal function"
30-sec chair stand test | Baseline, 8 weeks
  Score as 3-tier categories. Below Average; Average; Above Average. Sex- and age range-specific. "Below average" indicates a high risk of falls.
Functional reach test | Baseline, 8 weeks
  In standing, measures the distance between the length of an outstretched arm in a maximal forward reach; 10"/25 cm or greater: Low risk of falls; 6"/15cm to 10"/25cm: Risk of falling is 2x greater than normal; 6"/15cm or less: Risk of falling is 4x greater than normal; Unwilling to reach: Risk of falling is 8x greater than normal

CONTACTS AND LOCATIONS:
Locations (1):
- Michael.Ong@Cuhk.Edu.Hk, Hong Kong, NEW Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No